CLINICAL TRIAL: NCT01182649
Title: Randomized Comparison of Everolimus Eluting Stents and Sirolimus Eluting Stent in Patients With Coronary Artery Disease
Brief Title: Everolimus Stent in Patients With Coronary Artery Disease (CAD)
Acronym: RACES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: San Giuseppe Moscati Hospital (Other)
Responsible Party: EMILIO DI LORENZO MD PhD, DIVISION OF CARDIOLOGY AO MOSCATI
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOM_DES02
Record Dates: First submitted 2010-08-09; First posted 2010-08-17 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-05

CONDITIONS: Coronary Artery Disease; Coronary Atherosclerosis
Keywords: Drug Eluting Stents; Everolimus Eluting Stent; Coronary Angioplasty
MeSH Terms: conditions — Coronary Artery Disease | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EES Group (Experimental): Patients who received an everolimus eluting stent
  Interventions: Device: coronary stent
- SES Gruop (Active Comparator): Patients who received a sirolimus eluting stent
  Interventions: Device: stent

INTERVENTIONS:
Device: coronary stent — coronary angioplasty with stent implantation
  Other Names: XIENCE V drug eluting stent; Abbot Vascular USA
  Arms: EES Group
Device: stent — coronary angioplasty with stent implantation
  Other Names: CYPHER drug eluting stent; Johnson & Johnson USA
  Arms: SES Gruop

SUMMARY:
Aim of the study is to compare the everolimus eluting stent and sirolimus eluting stent in all comers PCI eligible patients

DETAILED DESCRIPTION:
Compared with the currently available first-generation drug-eluting stents (DES), second-generation DES have been designed with the goal of improving safety and efficacy. Everolimus, a sirolimus analogue, is released from a open cell, thin-strut, cobalt-chromium frame. A significant reduction in cardiac events was noted in patients with the everolimus-eluting stent compared with those who had a paclitaxel-eluting stent. Sirolimus eluting stent was the first available drug eluting stent and is the most tested. Therefore the investigators compared the safety and efficacy of the everolimus-eluting and sirolimus eluting stents in unselected patients in real world practice.

ELIGIBILITY:
Inclusion Criteria:

* All patients with coronary artery disease eligible for percutaneous coronary intervention (PCI)

Exclusion Criteria:

* Contraindication to dual antiplatelet therapy for 12 months
* Known allergy to sirolimus or everolimus
* Major surgical procedure planned within 1 month
* History, symptoms, or findings suggestive of aortic dissection.
* Participation in other trials
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Target Vessel Revascularization | 2 year
  Incidence of clinically driven target vessel revascularization at 2 year follow up

SECONDARY OUTCOMES:
cardiac death | 2 year
  incidence of death for cardiac causes at 2 year
non fatal myocardial infarction | 2 year
  incidence of non fatal Q or non Q wave reinfarction at 2 year
stent thrombosis | 2 year
  incidence of definite, probable or possible stent thrombosis at 2 year

CONTACTS AND LOCATIONS:
Overall Officials: EMILIO DI LORENZO, MD PhD, Principal Investigator — DIVISION OF CARDIOLOGY AORN MOSCATI AVELLINO ITALY
Locations (1):
- Division of Cardiology Aorn Moscati, Avellino, Italy

REFERENCES:
- [Background] Stone GW, Rizvi A, Newman W, Mastali K, Wang JC, Caputo R, Doostzadeh J, Cao S, Simonton CA, Sudhir K, Lansky AJ, Cutlip DE, Kereiakes DJ; SPIRIT IV Investigators. Everolimus-eluting versus paclitaxel-eluting stents in coronary artery disease. N Engl J Med. 2010 May 6;362(18):1663-74. doi: 10.1056/NEJMoa0910496. PMID 20445180
- [Background] Kedhi E, Joesoef KS, McFadden E, Wassing J, van Mieghem C, Goedhart D, Smits PC. Second-generation everolimus-eluting and paclitaxel-eluting stents in real-life practice (COMPARE): a randomised trial. Lancet. 2010 Jan 16;375(9710):201-9. doi: 10.1016/S0140-6736(09)62127-9. Epub 2010 Jan 7. PMID 20060578
- [Background] Caixeta A, Leon MB, Lansky AJ, Nikolsky E, Aoki J, Moses JW, Schofer J, Morice MC, Schampaert E, Kirtane AJ, Popma JJ, Parise H, Fahy M, Mehran R. 5-year clinical outcomes after sirolimus-eluting stent implantation insights from a patient-level pooled analysis of 4 randomized trials comparing sirolimus-eluting stents with bare-metal stents. J Am Coll Cardiol. 2009 Sep 1;54(10):894-902. doi: 10.1016/j.jacc.2009.04.077. PMID 19712798
- [Background] Di Lorenzo E, Sauro R, Varricchio A, Capasso M, Lanzillo T, Manganelli F, Mariello C, Siano F, Pagliuca MR, Stanco G, Rosato G, De Luca G. Benefits of drug-eluting stents as compared to bare metal stent in ST-segment elevation myocardial infarction: four year results of the PaclitAxel or Sirolimus-Eluting stent vs bare metal stent in primary angiOplasty (PASEO) randomized trial. Am Heart J. 2009 Oct;158(4):e43-50. doi: 10.1016/j.ahj.2009.03.016. PMID 19781402